CLINICAL TRIAL: NCT01025310
Title: Visual Stress of the Open Urban Environment
Status: Withdrawn | Type: Observational
Why Stopped: Administartive and technical problems
Sponsor: Meir Medical Center (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: 107-09
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2012-11

CONDITIONS: Visual Stress
Keywords: eye movements; saccades; visual; stress; search coil; environment; Saccadic eye movements; Urban environment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background and objectives: There is a general agreement that some types of urban environment could be the source of psychological stress as opposed to natural-relaxing environment. A number of aesthetical researches found out that the main cause for stress appearance can be explained by the complexity and order of the environment. There are also some indications that the stressing influence of the open environment can be measured by evaluating eye movements, in particular saccadic movements.

The objective of this study is to characterize eye movements - mainly saccades -while presenting visual material of different complexity and order and to evaluate the possible relationship between eye movements and parameters of psychological and physiological stress.

Methods: The research is based on systematic gradual experiments on healthy volunteers, who will be tested while viewing series of abstract figures and pictures of natural and urban areas with different level of complexity and order. Each figure or picture will be showed to subjects for 7 seconds. During the whole experimental session the investigators will measure:

1. Saccadic and other eye movements using the magnetic scleral search coil technique. The magnetic scleral search coil technique is the most sensitive and accurate technique used in modern ocular motor research for measuring horizontal, vertical and torsional eye movements. The coils are easy to apply and well tolerated over a wearing period of up to 45 minutes per recording session.
2. Heart rate pulse will be measured using a commercial pulse-meter.
3. Aesthetical evaluation: Following each figure or picture 7 seconds presentation; subjects will rate it in a scale from 1 (very relaxing) to 10 (very stressful).

Possible relationship between saccadic eye movements, heart rate and aesthetical rate will be analyzed using WIN 11 SPSS and MATLAB in statistically accepted ways.

Population: A total of about 60 healthy subjects aged 18-60 years old will be recruited for the study from students, faculty and staff of Tel Aviv University and of Meir Medical Center.

Criteria for inclusion: Healthy subject with normal vision

Criteria for exclusion: Eye disease such as corneal or scleral abrasion or disease, glaucoma, refractive errors greater than 2 diopters and concurrent medication with CNS-active agents.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Normal vision

Exclusion Criteria:

* Eye disease such as corneal or scleral abrasion or disease, glaucoma
* Refractive errors greater than 2 diopters
* Concurrent medication with CNS-active agents

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects aged 18-60 years old will be recruited for the study from students, faculty and staff of Tel Aviv University and of Meir Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos R Gordon, MD, DSc, Principal Investigator — Department of Neurology, Meir Medical Center, Kfar Saba, Israel
Locations (1):
- Department of Neurology, Kfar Saba, Kfar Saba, Israel